CLINICAL TRIAL: NCT03853928
Title: Multicenter, Randomized, Clinical Trial of Probiotics as Nutritional Support Versus Placebo in the Prevention of Hepatocellular Carcinoma in Cirrhosis
Brief Title: Probiotics in the Prevention of Hepatocellular Carcinoma in Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, Coordinator of Clinical Research Department, Austral University, Argentina
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-036
Record Dates: First submitted 2019-02-11; First posted 2019-02-26 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Microbiota; Hepatocellular Carcinoma; Cirrhosis
Keywords: Hepatocellular carcinoma; prevention; microbiome
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis | interventions — Probiotics; Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-controlled study of nutritional supplementation with probiotics to prevent the development of hepatocellular carcinoma in cirrhosis.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomized, double-blind, randomized controlled trial of probiotics versus placebo in patients with Child Pugh A-B cirrhosis at 3-year follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotics (Experimental): 50 ml bottle contains Lactobacillus casei 3.3 x 107 CFU / day, Lactobacillus plantarum 3.3 x 107 CFU / day, Streptococcus faecalis 3.3 x 107 CFU / day and Bifidobacterium brevis 1.0 x 106 CFU / day (BIOFLORA®, BIOSIDUS SA, Argentina) .
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): 5 ml orally every 12 hours for 10 consecutive days (Cycle, monthly). Duration of treatment Continuous, 1 cycle per month. Continuous treatment will be carried out from randomization to the development of the primary event or until the end of the study.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Each 50 ml bottle contains Lactobacillus casei 3.3 x 107 CFU / day, Lactobacillus plantarum 3.3 x 107 CFU / day, Streptococcus faecalis 3.3 x 107 CFU / day and Bifidobacterium brevis 1.0 x 106 CFU / day (BIOFLORA®, BIOSIDUS SA, Argentina) .
  Medication Reference intervention. Name of the active substance: Placebo. Administration way: Oral 5 ml orally every 12 hours for 10 consecutive days (Cycle, monthly)
  Likewise, both branches will explicitly request the non-consumption of alcohol and the consumption of a non-hypercaloric Mediterranean diet throughout the study for all patients in each branch (ANNEXIII).
  Other Names: Mediterranean diet

SUMMARY:
Background. The main risk factor for the development of hepatocellular carcinoma (HCC) is cirrhosis of any etiology, with an annual risk between 1 and 6%, being currently the leading cause of death in patients with cirrhosis and the third cause of death for cancer in the world. In our country there is little information about the incidence of HCC in this population. It has been shown that there is a change in the gut microbiome (set of genetic material of microorganisms that make up the intestinal bacterial flora) as the severity of the cirrhosis progresses. This change in the microbiome has been associated with clinical decompensation events of cirrhosis. However, there are no previous studies in the world that demonstrate an impact of the change of the microbiome in cirrhosis as a precursor to the development of HCC. Our team has compared the profile of the microbiome in patients with cirrhosis with and without HCC. We observed that patients with HCC present changes in the phylum Firmicutes, genus Fusobacterium and change in the bacteroides / prevotella ratio. This pattern was associated with a pro-inflammatory profile. In murine models, it has been postulated that modulation of the gut microbiome through the use of probiotics could have a clinical role in the prevention of HCC development.

This research project aims to answer the following question: in patients with cirrhosis, does the nutritional supplement with probiotics prevent HCC development? Objective: To compare the incidence of HCC through intervention with probiotics in cirrhosis.

Methods: A randomized, double-blind, placebo controlled trial of probiotics in patients with Child Pugh A-B cirrhosis at 3-year follow-up. Likewise, the type of microbiome found as a predictor of the risk of HCC development will be evaluated. It will include 280 patients, 140 in each branch. Basal blood and stool samples will be obtained and every 6 months. The typing and quantification of the microbiome in samples of fecal matter will be carried out by amplifying a specific region (V3-V4) of the bacterial 16s rRNA gene. Likewise, the presence of endotoxins (LPS) and cytokines (IL6, TNF alpha) in plasma will be determined to analyze the immune environment and the expression of the TLR4 receptor in mononuclear cells.

DETAILED DESCRIPTION:
Research question Does the modulation of gut microbiome with probiotics prevents the development of hepatocellular carcinoma in patients with cirrhosis? The aim of this study is to evaluate the efficacy of probiotics in reducing the incidence of hepatocellular carcinoma in patients with Child Pugh A-B cirrhosis with portal hypertension.

Methods Study design. Phase III interventional, multicenter, randomized, double-blind, placebo-controlled trial.

The following study will be carried out following CONSORT guidelines. Scenario and temporality. The study will be developed in Argentina including patient care centers with the following inclusion and exclusion criteria, from April 1/2019 (recruitment phase of 12 months) until the last enrolled patient completes the follow-up of 3 years from randomization.

Intervention. Test drug (s). Both probiotic and placebo will be presented in the same container, shape and color.

Name of the active substance Each 50 ml bottle contains Lactobacillus casei 3.3 x 107 CFU / day, Lactobacillus plantarum 3.3 x 107 CFU / day, Streptococcus faecalis 3.3 x 107 CFU / day and Bifidobacterium brevis 1.0 x 106 CFU / day (BIOFLORA®, BIOSIDUS SA, Argentina) .

Administration way: Oral 5 ml orally every 12 hours for 10 consecutive days per month. Duration of treatment: 2 cycles of continuous treatment per year during a 3-year period (6 cycles). Each cycle includes three months of treatment, followed by an off period of three months.

Reference intervention. Name of the active substance: Placebo. Administration way: Oral 5 ml orally every 12 hours for 10 consecutive days per month. Duration of treatment: 2 cycles of continuous treatment per year during a 3-year period (6 cycles). Each cycle includes three months of treatment, followed by an off period of three months.

**Likewise, both arms will explicitly request the non-consumption of alcohol and the consumption of a non-hypercaloric Mediterranean diet throughout the study for all patients.

Methodology. Patients who meet the aforementioned inclusion and exclusion criteria, and have successfully completed all screening tests, will be treated with the standard test or treatment medication according to clinical practice guidelines through a 1: 1 randomization scheme.

The randomization will be in stratified in blocks according to previously identified prognostic variables and in order to avoid potential confounding variables and or effect modifiers distributed by chance in an unbalanced way: Child Pugh score B and platelet count <100,000/mm3. The randomization will be carried out according to the assignment by means of numbers previously made by a blinded researcher and independent from clinical characteristics and contact with the patients. All numbers of the randomization will be stored in closed opaque envelopes and will be assigned consecutively according to the order of inclusion in the protocol.

*All the events developed, both primary and secondary throughout the study, will be evaluated by a blinded and independent committee from baseline variables and randomization allocation. Clinical events will be monitored and re-evaluated by this committee, which will consist of 3 investigators.

Exposure variables.

* Clinical Data
* Peripheral blood samples for the measurement of cytokines, LPS and expression of TLR 4.

  * Cytokines: The measurement of cytokines will be made from plasma of peripheral blood samples. The levels of the following cytokines will be quantified in pg/ml: IL-6, TNF-α and endotoxemia or bacterial lipopolysaccharide (LPS). The operators of this measurement will be blinded to any clinical, microbiome and treatment allocation. Samples to be obtained from each individual: two 10ml tubes of whole blood, one with EDTA (sodium ethylenediamine tetraacetate) and another without anticoagulant, to be used in routine laboratory studies and in the measurement of cytokines (IL6 and TNF alpha) and endotoxins (LPS). Quantification of plasma cytokines: Commercial reagents of enzyme-linked immunosorbent assay (ELISA) will be used to measure the levels of cytokines present in the plasmas of patients. The concentrations of TNF alpha and IL-6 will be measured with commercial reagents of eBioscience, affymetrix, or a similar commercial reagent available in the market, strictly following the instructions of the respective manufacturers. For the quantification of the cytokines, the curves will be made with the corresponding concentration standards.
  * Quantification of endotoxins in plasma or serum: Measurement of bacterial LPS will be performed by Limulus Amebocyte Lysate Assay (LAL), Biosafe Srl chromogenic endpoint reagent or similar, in parallel with the concentration curve of the standards. The manufacturer's instructions will be followed.
  * Expression of TLR 4 in peripheral blood mononuclear cells: the expression of TLR 4 in mononuclear cells will be quantified by real-time PCR technique, using specific primers.
  * Stool samples for gut microbiome evaluation.

    1. Method of Collection: A sample of spontaneous fecal stool will be collected at any time of the day in a supplied manifold avoiding contact with lavatory/odorless materials. Once the sample is collected, the appropriately capped collector will be placed inside a safety bag and inside a kit box. These samples will be stored frozen at -70º. Each fecal sample must be properly labeled. Later, samples will be aliquoted for final processing.
    2. Analysis: Fecal stools will be collected to analyze the gut microbiome using the PCR technique, Ilumina, analyzing the V3-V4 regions of 16sRNA at the biotechnology Institute of Rosario (INDEAR, Rosario, Argentina). The 16S ribosomal subunit of rRNA will be analyzed bacterial, amplifying using PCR method (20 cycles) and then a second round of amplification to incorporate multiplex adapters (Barcodes) (10 cycles). In each procedure, two measurements will be made to avoid amplification information biases. The massive sequencing will be carried out on an illumina MiSeq team from HERITAS institute (CIBIC + INDEAR) in 2x300 mode to finally obtain a minimum of 40,000 sequences per individual. The quality of the raw data will be evaluated by FastQC and the information of pair-ends of Illumina will be combined using PEAR (v0.9.10). The readings are then filtered by Q30 quality and the duplicates and PCR chimeras are eliminated using UCHIME. The filtered sequences will be clustered in Operational Taxonomic Units (OTUs) at 97% similarity with their own strategy implemented in QIIME (v1.91). The operators of this measurement will be blind to the clinical, microbiome, and primary event variables.
* The following measurements will be performed every 6 months in each subject enrolled until the end of the study or development of the primary event: weight and height, concomitant medication, complete physical examination, laboratory tests, Child Pugh score, abdominal ultrasound.
* Longitudinal sampling of gut microbiome and cytokines. A second cytokine measurement will be made from serum from peripheral blood and gut microbiome samples in fecal samples in all patients included in the study at the end of the first treatment cycle (3rd month since randomization or 12 weeks) and at the end of the study (last cycle) using the same methodology described above.

Adherence and Follow-up: All the patients will continue in the protocol until the development of the primary event or until the end of it, having completed a post-randomization follow-up of 3 years. Several measures will be carried out to reinforce adherence to treatment in both arms and strategies to avoid loss of follow-up. Adherence to treatment compliance will be defined in 80% of the tablets delivered for both arms.

Sample size calculation and statistical analysis: A two-tailed statistical value will be taken, α or type I error of 5% (p value <0.05) and a power or error type II or β of 0.20 (power of 80%). The risk of HCC in each arm will be compared using Cox regression analysis with Hazard Ratios (HR) and 95% confidence intervals and the number needed to treat to prevent a clinical outcome will be calculated, done according to the intention-to-treat principle. Since the cumulative incidence of HCC from previous data from the literature is 1-6% per year, a relative risk reduction of HCC development during a 3-year period in the intervention arm was estimated to be clinically relevant with a 30% relative difference, equivalent to a HR of 0.7. For each arm, a sample size of 140 subjects, with a total population to enroll of 280 patients, estimated number of primary events in 28.

All statistical analyzes will be carried out using STATA version 14.0.

Analysis of microbiome metadata. The bioinformatic analysis of the data will be done using a customized QIIME pipeline. For the estimation of differential abundance between the groups we use the DESeq2 package.

ELIGIBILITY:
Inclusion Criteria:

* signed Informed Consent (CI), obtained before carrying out any specific procedure of the study
* Clinical or histological diagnosis of cirrhosis
* Child Pugh A or B
* Presence of clinical signs of portal hypertension: esophagogastric varices or hypertensive gastropathy or edematous ascitic syndrome or encephalopathy.

Exclusion Criteria:

* History of hepatocellular carcinoma prior to randomization
* Solid organ transplant.
* Immunosuppressive treatment.
* Previous treatment (during the last 6 months prior to the inclusion of the study) or current with pre or probiotics.
* Current antibiotic treatment for any reason.
* Active alcoholism: alcohol consumption in the last 3 months prior to randomization.
* History or current history of other neoplasms.
* Major surgical intervention or serious traumatic injury in the 28 days prior to randomization.
* Unstable angina (angina symptoms at rest, recently started angina, or within the last 3 months of randomization) or myocardial infarction in the 6 months prior to randomization.
* Uncontrolled cardiac arrhythmia, valvular heart disease.
* Infection grade> 2 in progress, according to the NCA CTCAE criteria, version 4.0.
* Inflammatory bowel disease including ulcerative colitis and Crohn's disease.
* Celiac Disease.
* Diarrhea secondary to any germ or commensal, including Clostridium difficile diarrhea within 6 months prior to randomization.
* Any malabsorption disorder.
* Chronic renal failure with hemodialysis requirement.
* Known hypersensitivity to any of the study drugs, to the study drug classes or to the excipients of its formulation.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients developing Hepatocellular carcinoma | 3 years of follow-up
  The aim of this study is to evaluate the efficacy of probiotics in patients with Child Pugh A-B cirrhosis in reducing the incidence of hepatocellular carcinoma.
  The main measure of effectiveness in this study is the development of Hepatocarcinoma.

SECONDARY OUTCOMES:
Description of type of gut microbiome found in cirrhosis with or without treatment with probiotics. | Three year period
  Evaluate intestinal microbiome changes and analyze their association with the development of HCC.
Analyze the immunological context found in cirrhosis with or without treatment with probiotics. | Three year period
  Analyze the presence of an immune environment that contributes to the development of this cancer.
Number of Liver decompensation events in cirrhosis with or without treatment with probiotics. | Three year period
  Study the development of new complications of portal hypertension with the use of probiotics: ascites, portosystemic encephalopathy and variceal bleeding.
Adverse events found in cirrhosis with or without treatment with probiotics. | Three year period
  Analyze adverse events related to the use of probiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Piñero, MD, MSCE, Principal Investigator — Austral University, Argentina

IPD SHARING:
Plan to Share IPD: No